CLINICAL TRIAL: NCT02879448
Title: AMPLATZER™ Amulet™ Left Atrial Appendage Occluder Randomized Controlled Trial
Brief Title: AMPLATZER™ Amulet™ LAA Occluder Trial
Acronym: Amulet IDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SJM-CIP-10114
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Non-valvular atrial fibrillation; Left Atrial Appendage
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amulet (Experimental): Amulet left atrial appendage occluder
  Interventions: Device: Amulet Left Atrial Appendage Occluder
- WATCHMAN (Control) (Active Comparator): WATCHMAN left atrial appendage closure device
  Interventions: Device: WATCHMAN Left Atrial Appendage Closure

INTERVENTIONS:
Device: Amulet Left Atrial Appendage Occluder — Transcatheter left atrial appendage closure
  Arms: Amulet
Device: WATCHMAN Left Atrial Appendage Closure — Transcatheter left atrial appendage closure
  Arms: WATCHMAN (Control)

SUMMARY:
The Amulet™ device will be evaluated for safety and efficacy by demonstrating its performance is non-inferior to the commercially available WATCHMAN® left atrial appendage closure device in patients with non-valvular atrial fibrillation. Patients who are eligible for the trial will be randomized to receive either the Amulet device or the WATCHMAN device and will be followed for 5 years after device implant.

DETAILED DESCRIPTION:
The Amulet IDE trial is a prospective, randomized, multi-center active control worldwide trial, designed to evaluate the safety and effectiveness of the AMPLATZER™ Amulet™ Left Atrial Appendage Occluder. Subjects will be randomized in a 1:1 ratio between the Amulet left atrial appendage (LAA) occlusion device (treatment) or a Boston Scientific WATCHMAN® LAA closure device (Control). The trial will be conducted at up to 150 sites worldwide. All enrolled subjects will follow the protocol-required tests and assessments at each scheduled follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF) and the patient has not been diagnosed with rheumatic mitral valvular heart disease
3. At high risk of stroke or systemic embolism defined as CHADS2 score ≥ 2 or a CHA2DS2-VASc score of ≥ 3
4. Has an appropriate rationale to seek an alternative to warfarin or other anticoagulation medication
5. Deemed by investigator to be suitable for short term warfarin therapy but deemed unable to take long term oral anticoagulation, following the conclusion of shared decision making (see inclusion criteria #6)
6. Deemed suitable for LAA closure by a multidisciplinary team of medical professionals (including an independent non-interventional physician) involved in the formal and shared decision- making process, and by use of an evidence-based decision tool on oral anticoagulation (final determination must be documented in the subject's medical record)
7. Able to comply with the required medication regimen post-device implant
8. Able to understand and willing to provide written informed consent to participate in the trial
9. Able and willing to return for required follow-up visits and examinations

Exclusion Criteria:

1. Requires long-term oral anticoagulation therapy for a condition other than atrial fibrillation
2. Contraindicated for or allergic to aspirin, clopidogrel, or warfarin use
3. Indicated for chronic P2Y12 platelet therapy inhibitor
4. Is considered at high risk for general anesthesia, in the opinion of the investigator, and/or based on past adverse reaction(s) requiring medical intervention or which resulted in prolongation of hospital stay (criterion is only applicable where general anesthesia is planned for the study procedure).
5. Has undergone atrial septal defect (ASD) repair or has an ASD closure device present
6. Has undergone patent foramen ovale (PFO) repair or has a PFO closure device implanted
7. Implanted with a mechanical valve prosthesis
8. Has any of the customary contraindications for a percutaneous catheterization procedure (e.g. subject is too small to accommodate the transesophageal echocardiogram (TEE/TOE) probe or required catheters, or subject has active infection or bleeding disorder)
9. Stroke or transient ischemic attack (TIA) within 90 days prior to randomization or implant procedure (as applicable)
10. Underwent any cardiac or non-cardiac intervention or surgery within 30 days prior to randomization, or intervention or surgery is planned within 60 days after implant procedure (e.g. cardioversion, ablation, cataract surgery, etc.)
11. Myocardial infarction (MI) within 90 days prior to randomization
12. New York Heart Association Class IV Congestive Heart Failure
13. Left ventricular ejection Fraction (LVEF) ≤30%
14. Symptomatic carotid artery disease (defined as >50% stenosis with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is <50% stenosis
15. Reversible cause of AF (i.e. secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
16. History of idiopathic or recurrent venous thromboembolism
17. Left atrial appendage is obliterated or surgically ligated
18. Thrombocytopenia or anemia requiring transfusions
19. Hypersensitivity to any portion of the device material or individual components of either the Amulet or Boston Scientific LAA closure device (e.g. nickel allergy)
20. Actively enrolled or plans to enroll in a concurrent clinical study in which the active treatment arm may confound the results of this trial
21. Subject is pregnant or pregnancy is planned during the course of the investigation
22. Active endocarditis or other infection producing bacteremia
23. Subject has had a transient case of AF (i.e. never previously detected, provoked/induced by surgical or catheter manipulations, etc.)
24. Subjects with severe renal failure (estimated glomerular filtration rate <30ml/min/1.73m²)
25. Subject whose life expectancy is less than 2 years
26. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical trial or to comply with follow up requirements, or impact the scientific soundness of the clinical trial results.

Echocardiographic Exclusion Criteria:

1. Intracardiac thrombus visualized by echocardiographic imaging
2. Existing circumferential pericardial effusion >2mm
3. Significant mitral valve stenosis (i.e. mitral valve area <1.5 cm^2)
4. High risk PFO, defined as an atrial septal aneurysm (excursion > 15mm or length ≥ 15mm; excursion defined as maximal protrusion of the atrial septal aneurysm [ASA] beyond the plane of the atrial septum) or large shunt (early, within 3 beats and/or substantial passage of bubbles i.e. ≥ 20)
5. Complex atheroma with mobile plaque of the descending aorta and/or aortic arch
6. Cardiac tumor
7. LAA anatomy cannot accommodate either a Boston Scientific LAA closure device or Amulet device, as per manufacturer's Instructions for Use (IFU). (i.e. the LAA anatomy and sizing must be appropriate for both devices in order to be enrolled in the trial. This is applicable to all roll-in and randomized subjects).
8. Placement of the device would interfere with any intracardiac or intravascular structure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1878 (Actual)
Dates: Start 2016-08-24; Primary Completion 2020-12-07 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Study Chair — University of Kansas; David Thaler, MD, PhD, Study Chair — The Comprehensive Stroke Center at Tufts Medical Center; Stephan Windecker, MD, PhD, Study Chair — Inselspital, University of Bern
Locations (115):
- United States (85):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Scripps Health, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC University Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - University of California - Davis Medical Center, Sacramento, California
  - Mercy Medical Group - Cardiology, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - Pacific Heart Institute, Santa Monica, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Bradenton Cardiology Center, Bradenton, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Watson Clinic Center, Lakeland, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - VA Medical Center Minneapolis, Minneapolis, Minnesota
  - St. Cloud Hospital (Central MN Heart Clinic), Saint Cloud, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Albany Medical Center, Albany, New York
  - Winthrop-University Hospital, Mineola, New York
  - New York University Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian/Columbia University Medical Center, New York, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt Heart Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Austin Heart, Austin, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin
- Australia (4):
  - Specialist Cardiology, Wahroonga, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - St. Andrew's Hospital, Adelaide, South Australia
  - HeartCare St John of God Wexford Medical Centre, Murdoch, Western Australia
- Canada (2):
  - Vancouver General Hospital (U of BC), Vancouver, British Columbia
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- Nemocnice Na Homolce, Prague, Central Bohemia, Czechia
- Denmark (2):
  - Skejby University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- Germany (12):
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen, Bad-wur
  - Klinikum Coburg GmbH, Coburg, Bavaria
  - Internistisches Klinikum München SUD, Munich, Bavaria
  - Cardioangiologisches Centrum am Bethanien Krankenhaus, Frankfurt am Main, Hesse
  - CardioVaskuläres Centrum St. Katharinen, Frankfurt am Main, Hesse
  - Evangelisches Krankenhaus Bielefeld, Bielefeld, North Rhine
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf, North Rhine
  - Elisabeth-Krankenhaus Essen GmbH, Essen, North Rhin
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - Asklepios Klinik St. Georg, Hamburg
- Ospedale San Raffaele - Aritmologia, Milan, Lombard, Italy
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands
- Santa Maria Hospital, Lisbon, Lisbon District, Portugal
- Spain (5):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital General Juan Ramon Jimenez, Huelva, Andalu
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Catalonia
  - Clínica Universidad de Navarra, Pamplona, Navarre
- Center Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen-Kudsk JE, Schmidt B, Windecker S, Shah N, Gray W, Ellis CR, Koulogiannis K, Anderson JA, Gage R, Lakkireddy D. Characterization and Clinical Outcomes of High-Risk Device-Related Thrombus in the Amulet IDE Trial. JACC Clin Electrophysiol. 2025 Jul;11(7):1543-1554. doi: 10.1016/j.jacep.2025.02.016. Epub 2025 Apr 9. PMID 40208159
- [Derived] Lakkireddy D, Ellis CR, Thaler D, Swarup V, Gambhir A, Hermiller J, Nielsen-Kudsk JE, Worthley S, Nair D, Schmidt B, Horton R, Gupta N, Anderson JA, Zhao H, Alkhouli M, Windecker S. 5-Year Results From the AMPLATZER Amulet Left Atrial Appendage Occluder Randomized Controlled Trial. J Am Coll Cardiol. 2025 Mar 25;85(11):1141-1153. doi: 10.1016/j.jacc.2024.10.101. Epub 2024 Nov 18. PMID 39570242
- [Derived] Lakkireddy D, Thaler D, Ellis CR, Swarup V, Gambhir A, Hermiller J, Nielsen-Kudsk JE, Worthley S, Nair D, Schmidt B, Horton R, Gupta N, Anderson JA, Gage R, Alkhouli M, Windecker S. 3-Year Outcomes From the Amplatzer Amulet Left Atrial Appendage Occluder Randomized Controlled Trial (Amulet IDE). JACC Cardiovasc Interv. 2023 Aug 14;16(15):1902-1913. doi: 10.1016/j.jcin.2023.06.022. PMID 37587599
- [Derived] Lakkireddy D, Nielsen-Kudsk JE, Windecker S, Thaler D, Price MJ, Gambhir A, Gupta N, Koulogiannis K, Marcoff L, Mediratta A, Anderson JA, Gage R, Ellis CR. Mechanisms, predictors, and evolution of severe peri-device leaks with two different left atrial appendage occluders. Europace. 2023 Aug 2;25(9):euad237. doi: 10.1093/europace/euad237. PMID 37584233
- [Derived] Schmidt B, Nielsen-Kudsk JE, Ellis CR, Thaler D, Sabir SA, Gambhir A, Landmesser U, Shah N, Gray W, Swarup V, Lim DS, Koulogiannis K, Anderson JA, Gage R, Lakkireddy D. Incidence, Predictors, and Clinical Outcomes of Device-Related Thrombus in the Amulet IDE Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):96-107. doi: 10.1016/j.jacep.2022.07.014. Epub 2022 Sep 28. PMID 36697204
- [Derived] Alkhouli M, Russo AM, Thaler D, Windecker S, Anderson JA, Gage R, Lakkireddy D. Sex Differences in Safety and Effectiveness of LAAO: Insights From the Amulet IDE Trial. JACC Cardiovasc Interv. 2022 Nov 14;15(21):2143-2155. doi: 10.1016/j.jcin.2022.06.037. Epub 2022 Oct 12. PMID 36357018
- [Derived] Price MJ, Ellis CR, Nielsen-Kudsk JE, Thaler D, Gupta N, Koulogiannis K, Anderson JA, Gage R, Lakkireddy D. Peridevice Leak After Transcatheter Left Atrial Appendage Occlusion: An Analysis of the Amulet IDE Trial. JACC Cardiovasc Interv. 2022 Nov 14;15(21):2127-2138. doi: 10.1016/j.jcin.2022.09.001. PMID 36357016
- [Derived] Lakkireddy D, Thaler D, Ellis CR, Swarup V, Sondergaard L, Carroll J, Gold MR, Hermiller J, Diener HC, Schmidt B, MacDonald L, Mansour M, Maini B, O'Brien L, Windecker S. Amplatzer Amulet Left Atrial Appendage Occluder Versus Watchman Device for Stroke Prophylaxis (Amulet IDE): A Randomized, Controlled Trial. Circulation. 2021 Nov 9;144(19):1543-1552. doi: 10.1161/CIRCULATIONAHA.121.057063. Epub 2021 Aug 30. PMID 34459659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2079 subjects were enrolled at 115 investigational centers and Amulet IDE trial included 2079 subjects with 1878 Randomized subjects (934 in the Amulet group and 944 in the Watchman group) and 201 roll-in subjects.
Pre-assignment Details: Of the 2592 subjects who consented initially, 513 subjects did not enroll in the Amulet IDE trial due to screen failures, withdrawal of consent, and other reasons. Hence, the actual enrollment was 1878 Randomized subjects and 201 roll-in subjects.
Period: Overall Study
Arm/Group | Amulet | WATCHMAN (Control)
Started | 934 | 944
Completed | 610 | 562
Not Completed | 324 | 382
Not completed — Death | 251 | 263
Not completed — Lost to Follow-up | 23 | 28
Not completed — Withdrawal by Subject | 42 | 79
Not completed — Other Reasons | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amulet | WATCHMAN (Control) | Total
Number analyzed (Participants) | 934 | 944 | 1878
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (7.6) | 75.1 (7.6) | 75.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 365 | 750
  Male | 549 | 579 | 1128
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were identified in both Race and Ethnicity
  Participants
    White | 838 | 851 | 1689
    Black or African American | 21 | 20 | 41
    Asian | 4 | 7 | 11
    American Indian or Alaska Native | 4 | 2 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
    Other | 10 | 9 | 19
    Declined or Unable to Disclose Due to Local Regulation | 57 | 52 | 109
    Hispanic or Latino | 26 | 35 | 61
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 7
  Europe | 102 | 101 | 203
  United States | 792 | 806 | 1598
  Australia | 36 | 34 | 70
History of major or minor bleeding [Count of Participants; unit: Participants] | 515 | 503 | 1018

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Composite Endpoint Rate of Procedure-related Complications, or All-cause Death or Major Bleeding (Defined as Type 3 or Greater Based on the Bleeding Academic Research Consortium (BARC) Definition) (Non-inferiority Analysis)
Description: Procedure related complications are adverse events adjudicated by the Clinical Events Committee (CEC), as procedure related and requiring either invasive surgical or percutaneous intervention.
  All-cause deaths (cardiovascular or non-cardiovascular) were assessed.
  Major Bleeding
  * Type 3a:
    * Any transfusion with overt bleeding
    * Overt bleeding+Hb drop of ≥ 3 to < 5 g/dL (provided Hb drop is related to bleed)
  * Type 3b:
    * Overt bleeding+Hb drop ≥ 5 g/dL (provided Hb drop is related to bleed)
    * Cardiac tamponade
    * Bleeding requiring surgical intervention for (Watchman)
    * Bleeding requiring intravenous vasoactive drugs
  * Type 3c:
    * Intracranial hemorrhage including subdural hemorrhages
    * Subcategories confirmed by autopsy/imaging/lumbar puncture
    * Intraocular bleed compromising vision
  * Type 5a: Probably fatal bleeding
  * Type 5b: Definite fatal bleeding
Time Frame: At 12-months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 903 | 896
Percentage of participants | 14.5 | 14.7
Statistical Analysis 1: Comparison: WATCHMAN (Control); The following hypothesis was tested: H0: p1(Amulet) - p1 (Watchman) ≥ Δ1 H1: p1(Amulet) - p1(Watchman) < Δ1; where Δ1 is the absolute value of the non-inferiority margin for the safety endpoint and p1 is the probability of a primary safety endpoint event; Test type: Non-Inferiority — The non-inferiority margin was developed based on reported rates for other devices. Therefore, the expected rate of the safety endpoint was assumed to be 15%. A non-inferiority margin of 5.8% represents a relative risk of 1.39; p = 0.0002, Kaplan-Meier estimate

2. Primary Outcome: Primary Effectiveness Endpoint: Composite Rate of Ischemic Stroke or Systemic Embolism (Non-inferiority Analysis)
Description: Ischemic Stroke: An acute symptomatic episode of focal cerebral, spinal, or retinal dysfunction caused by an infarction of central nervous system tissue.
  Systemic Embolism: Acute vascular insufficiency or occlusion of the extremities or any non-central nervous system (non-CNS) organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (e.g. trauma, atherosclerosis, or instrumentation). When there is presence of prior peripheral artery disease, angiographic or surgical or autopsy evidence is required to show abrupt arterial occlusion.
Time Frame: At 18-months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 934 | 944
Percentage of participants | 2.8 | 2.8
Statistical Analysis 1: Comparison: WATCHMAN (Control); The following hypothesis was tested: H0: p2(Amulet) - p2(Watchman) ≥ Δ2 H1: p2(Amulet) - p2(Watchman) < Δ2; where Δ2 is the absolute value of the non-inferiority margin for the effectiveness endpoint and p2 is the probability of a subject experiencing a primary effectiveness endpoint event; Test type: Non-Inferiority — The non-inferiority margin for this endpoint was developed based on the reported rates of ischemic stroke or systemic embolism for the Watchman. The 18-month rate of ischemic stroke or systemic embolism for the Watchman device has been reported in the literature as 4.2%. A non-inferiority margin of 3.2%, which represents a relative risk of 1.76, ensured that the rate observed was at most twice the rate expected with oral anticoagulant therapy; p < 0.0001, Kaplan-Meier estimate

3. Primary Outcome: Mechanism of Action Primary Endpoint: Rate of Device Closure, by the Echocardiography Core Lab (Non-inferiority Analysis)
Description: Device closure (defined as residual jet around the device ≤ 5 mm) at the 45-day visit documented by transesophageal echocardiogram (TEE/TOE) defined by Doppler flow was assessed.
Time Frame: At 45-days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 801 | 792
Percentage of participants | 98.9 | 96.8
Statistical Analysis 1: Comparison: WATCHMAN (Control); The following hypothesis was tested: H0: p3(Amulet) - p3(Watchman) ≤ -Δ3 H1: p3(Amulet) - p3(Watchman) > -Δ3; where Δ3 is the absolute value of the non-inferiority margin and p3 is the 45-day closure probability; Test type: Non-Inferiority — The non-inferiority margin for this endpoint was developed based on the reported closure rate for the Watchman device. The rate of device closure for the Watchman device has been reported in the literature as 95% (i.e., 5% had a residual jet > 5mm). A non-inferiority margin of -3%, which represents a relative risk of 1.60, allows for trial to trial variability and implanter learning associated with implantation of a new device (Amulet); p < 0.0001, Farrington Manning test

4. Secondary Outcome: Composite Rate of All Stroke, Systemic Embolism, or Cardiovascular/Unexplained Death (Non-inferiority Analysis)
Description: Stroke: An acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.
  Systemic Embolism: Acute vascular insufficiency/occlusion of the extremities/any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (trauma/atherosclerosis/instrumentation). When there is presence of prior peripheral artery disease, angiographic/surgical/autopsy evidence is required to show abrupt arterial occlusion.
  Cardiovascular/unexplained death includes:
  * Death due to proximate cardiac cause
  * Death caused by non-coronary/non-CNS vascular conditions
  * Death from vascular CNS causes
  * All procedure-related deaths
  * Sudden/unwitnessed death
  * Death of unknown cause
Time Frame: At 18-months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 915 | 916
Percentage of participants | 5.6 | 7.7
Statistical Analysis 1: Comparison: WATCHMAN (Control); Test type: Non-Inferiority — The following hypothesis was tested: H1: p4(Amulet) - p4(Watchman) < 4.5%; p < 0.0001, Kaplan-Meier estimate

5. Secondary Outcome: Rate of Major Bleeding (Superiority Analysis)
Description: Major bleeding rate defined as Type 3 or greater based on the Bleeding Academic Research Consortium (BARC) definition was assessed
  * Type 3a:
    * Any transfusion with overt bleeding
    * Overt bleeding+Hb drop of ≥ 3 to < 5 g/dL (provided Hb drop is related to bleed)
  * Type 3b:
    * Overt bleeding+Hb drop ≥ 5 g/dL (provided Hb drop is related to bleed)
    * Cardiac tamponade
    * Bleeding requiring surgical intervention for (Watchman)
    * Bleeding requiring intravenous vasoactive drugs
  * Type 3c:
    * Intracranial hemorrhage including subdural hemorrhages
    * Subcategories confirmed by autopsy/imaging/lumbar puncture
    * Intraocular bleed compromising vision
  * Type 5a: Probably fatal bleeding: bleeding that is clinically suspicious as the cause of death, but the bleeding is not directly observed and there is no autopsy or confirmatory imaging
  * Type 5b: Definite fatal bleeding: bleeding that is directly observed or confirmed on autopsy
Time Frame: At 18-months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 917 | 916
Percentage of participants | 11.6 | 12.3
Statistical Analysis 1: Comparison: WATCHMAN (Control); Test type: Superiority — The following hypothesis was tested: H1: p5(Amulet) - p5(Watchman) < 0; p = 0.3229, Kaplan-Meier estimate

6. Secondary Outcome: Superiority Test of Primary Safety Endpoint: Composite Endpoint Rate of Procedure-related Complications, or All-cause Death or Major Bleeding (Defined as Type 3 or Greater Based on the Bleeding Academic Research Consortium (BARC) Definition)
Description: as for outcome 1
Time Frame: At 12-months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 903 | 896
percentage of participants | 14.5 | 14.7
Statistical Analysis 1: Comparison: WATCHMAN (Control); Test type: Superiority — The following hypothesis was tested: H1: p1(Amulet) - p1(Watchman) < 0; p = 0.4660, Kaplan-Meier estimate

7. Secondary Outcome: Superiority Test of Primary Effectiveness Endpoint: Composite Rate of Ischemic Stroke or Systemic Embolism
Description: as for outcome 2
Time Frame: At 18-months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 934 | 944
Percentage of participants | 2.8 | 2.8
Statistical Analysis 1: Comparison: WATCHMAN (Control); Test type: Superiority — The following hypothesis was tested: H1: p2(Amulet) - p2(Watchman) < 0; p = 0.5017, Kaplan-Meier estimate

8. Secondary Outcome: Superiority Test of Primary Mechanism of Action Endpoint: Rate of Device Closure, by the Echocardiography Core Lab
Description: as for outcome 3
Time Frame: At 45-days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 801 | 792
Percentage of participants | 98.9 | 96.8
Statistical Analysis 1: Comparison: WATCHMAN (Control); Test type: Superiority — The following hypothesis was tested: H1: p3(Amulet) - p3(Watchman) > 0; p = 0.0025, Farrington Manning test

9. Post Hoc Outcome: Composite Rate of Ischemic Stroke and Systemic Embolism
Description: Ischemic Stroke is defined as an acute symptomatic episode of focal cerebral, spinal, or retinal dysfunction caused by an infarction of central nervous system tissue and Systemic Embolism is define as Acute vascular insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (e.g. trauma, atherosclerosis, or instrumentation). When there is presence of prior peripheral artery disease, angiographic or surgical or autopsy evidence is required to show abrupt arterial occlusion.
Time Frame: 5 Years
Population: Analysis included subjects who underwent an implant attempt regardless of the device attempted or implanted.
Measure: Number; unit: percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 917 | 916
percentage of participants | 7.4 | 7.1

10. Post Hoc Outcome: Composite Rate of Stroke, Systemic Embolism, or CV/Unexplained Death
Description: Stroke: An acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.
  Systemic Embolism: Acute vascular insufficiency/occlusion of the extremities/any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (trauma/atherosclerosis/instrumentation). When there is presence of prior peripheral artery disease, angiographic/surgical/autopsy evidence is required to show abrupt arterial occlusion.
  Cardiovascular/unexplained death includes:
  Death due to proximate cardiac cause Death caused by non-coronary/non-CNS vascular conditions Death from vascular CNS causes All procedure-related deaths Sudden/unwitnessed death Death of unknown cause
Time Frame: 5 Years
Population: Analysis included subjects who underwent an implant attempt regardless of the device attempted or implanted.
Measure: Number; unit: percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 917 | 916
percentage of participants | 20.3 | 20.7

11. Post Hoc Outcome: Rate of Major Bleeding
Description: Major bleeding:
  Type 3a: Any transfusion with overt bleeding. Overt bleeding plus a hemoglobin drop of ≥ 3 to < 5 g/dL.
  Type 3b: Overt bleeding plus hemoglobin drop ≥ 5 g/dL. Cardiac tamponade. Bleeding requiring surgical intervention for Watchman (excluding dental/nasal/skin/ hemorrhoid). Bleeding requiring intravenous vasoactive drugs.
  Type 3c:Intracranial hemorrhage including subdural hemorrhages (does not include microbleeds or hemorrhagic transformation, does include intraspinal). Subcategories confirmed by autopsy or imaging or lumbar puncture. Intraocular bleed compromising vision.
  Type 5a: Probably fatal bleeding: bleeding that is clinically suspicious as the cause of death, but the bleeding is not directly observed and there is no autopsy or confirmatory imaging.
  Type 5b: Definite fatal bleeding: bleeding that is directly observed (by either clinical specimen) or confirmed on autopsy.
Time Frame: 5 Years
Population: Analysis included subjects who underwent an implant attempt regardless of the device attempted or implanted.
Measure: Number; unit: percentage of participants
Arm/Group | Amulet | WATCHMAN (Control)
Number analyzed (Participants) | 917 | 916
percentage of participants | 20.1 | 20.0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Amulet | WATCHMAN (Control)
All-Cause Mortality (participants affected / at risk) | 251/934 | 263/944
Serious Adverse Events (participants affected / at risk) | 542/934 | 535/944
Other Adverse Events (participants affected / at risk) | 293/934 | 266/944
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amulet (N=934) | WATCHMAN (Control) (N=944)
Anemias (Blood and lymphatic system disorders) | 33 | 25
Aplastic Anemia/Hypoplastic Anemia (Blood and lymphatic system disorders) | 2 | 2
Iron-Deficiency Anemia (Blood and lymphatic system disorders) | 0 | 3
Aortic Valve Insufficiency/Aortic Valve Regurgitation/Valvular Regurgitation Aortic Valve (Cardiac disorders) | 1 | 1
High Grade Block/Advanced AV Block (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation: Tricuspid Valve (Cardiac disorders) | 2 | 2
AV Block (Cardiac disorders) | 1 | 0
Acute Pulmonary Edema (Cardiac disorders) | 2 | 0
Angina Pectoris (Cardiac disorders) | 1 | 5
Anterior Myocardial Infarction (Cardiac disorders) | 27 | 22
Aortic Aneurysms (Cardiac disorders) | 3 | 1
Aortic Dissection (Cardiac disorders) | 1 | 1
Aortic Valve Stenosis (Cardiac disorders) | 7 | 4
Asystole (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 4 | 1
Cardiac Arrest (Cardiac disorders) | 36 | 39
Cardiac Perforation (Cardiac disorders) | 1 | 1
Cardiac Thrombus (Cardiac disorders) | 1 | 1
Cardiogenic Shock (Cardiac disorders) | 4 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Chest Pain (Cardiac disorders) | 13 | 20
Congestive Heart Failure (Cardiac disorders) | 113 | 105
Constrictive Pericarditis (Cardiac disorders) | 1 | 0
Cor Pulmonale (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 11 | 13
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Dyspnea (Cardiac disorders) | 4 | 3
Inferior Myocardial Infarction (Cardiac disorders) | 2 | 0
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 9 | 5
Myocardial Infarction (Cardiac disorders) | 1 | 0
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 17 | 7
Pericardial Tamponade (Cardiac disorders) | 18 | 14
Pericarditis (Cardiac disorders) | 8 | 2
Perivalvular Leak (Cardiac disorders) | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 8 | 6
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 7 | 4
Sinus Node Dysfunction (Cardiac disorders) | 1 | 1
Supravalvular Aortic Stenosis (Cardiac disorders) | 1 | 0
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 | 2
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 2 | 3
Unstable Angina (Cardiac disorders) | 3 | 5
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 4 | 1
Eye Bleed (Eye disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Acute Peritonitis (Gastrointestinal disorders) | 1 | 1
Bowel Obstruction (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Emesis/Vomiting (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal Bleeding (Gastrointestinal disorders) | 98 | 99
Hemorrhoids/Piles (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Hemiparesis/Weakness (General disorders) | 1 | 0
Tingling (General disorders) | 0 | 1
Weakness (General disorders) | 6 | 4
Damage or Movement of ICD Leads Requiring Revisions (General disorders) | 1 | 0
Drug Side Effect (General disorders) | 1 | 0
Failure to Thrive (General disorders) | 7 | 9
Fatigue/Generalized Fatigue (General disorders) | 3 | 1
Fever (General disorders) | 1 | 4
Multiple Organ Failure (General disorders) | 17 | 16
Neck Pain (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 3 | 3
Other (General disorders) | 25 | 25
Choledocholithiaisis (Hepatobiliary disorders) | 1 | 0
Ascites (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Choledocholithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic and Biliary Disorders (Hepatobiliary disorders) | 3 | 3
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (Infections and infestations) | 1 | 1
Bacterial Infections of the Skin (Infections and infestations) | 0 | 1
Subacute Bacterial Endocarditis (SBE) (Infections and infestations) | 1 | 0
Acute Bacterial Endocarditis (ABE) (Infections and infestations) | 2 | 0
Bacteremia (Infections and infestations) | 1 | 1
Bacterial Infections (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Chlamydial Pneumonia (Infections and infestations) | 1 | 0
Infected Cyst (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 24
Respiratory Syncytial Virus Infection (RSV) (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 22 | 18
Septicemia (Infections and infestations) | 1 | 0
Urinary Tract Infections (Infections and infestations) | 6 | 7
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Air Embolus (Injury, poisoning and procedural complications) | 2 | 2
Closed Head Injury (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Epidural Hematomas (Injury, poisoning and procedural complications) | 1 | 0
Esophageal Laceration and Rupture (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 7 | 13
Hemothorax (Injury, poisoning and procedural complications) | 4 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Trauma (Injury, poisoning and procedural complications) | 29 | 29
VASC Bleeding (Injury, poisoning and procedural complications) | 1 | 3
VASC Hematoma (Injury, poisoning and procedural complications) | 3 | 8
VASC Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 4
VASC Vessel Perforation (Injury, poisoning and procedural complications) | 1 | 1
Abnormal Coagulation Parameter (Investigations) | 0 | 4
Abnormal Lab Value (Investigations) | 2 | 4
EKG Abnormalities (Investigations) | 1 | 0
Echo Finding (Investigations) | 0 | 1
Poor Nutrition (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Edema (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 | 28
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukemias (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Edema (Nervous system disorders) | 1 | 0
Dysarthria/Slurred Speech (Nervous system disorders) | 0 | 1
Facial Paresis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracerebral Haemorrhage (Nervous system disorders) | 9 | 6
Intraventricular Haemorrhage (Nervous system disorders) | 1 | 0
Ischemic Stroke (Nervous system disorders) | 57 | 53
Stroke (Nervous system disorders) | 2 | 1
Unmasking Old Stroke Symptoms (Nervous system disorders) | 1 | 0
Visual Disturbance (Nervous system disorders) | 1 | 0
Acute Subdural Hematoma (Nervous system disorders) | 3 | 1
Altered Sensorium (Nervous system disorders) | 0 | 2
Ataxia (Nervous system disorders) | 0 | 1
Bells Palsy (Nervous system disorders) | 0 | 1
Blurred Vision (Nervous system disorders) | 0 | 1
Cerebral Aneurysm (Nervous system disorders) | 1 | 1
Concussion (Nervous system disorders) | 0 | 1
Delirium (Nervous system disorders) | 2 | 3
Dementia (Nervous system disorders) | 5 | 9
Dizziness (Nervous system disorders) | 6 | 2
Dysphasia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 22 | 24
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0
Microhemorrhage (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Neuralgic Facial Pain (Nervous system disorders) | 1 | 0
New and Different Onset of Migraine Symptoms (Nervous system disorders) | 2 | 0
Numbness (Nervous system disorders) | 1 | 0
Parkinson's Disease (Nervous system disorders) | 4 | 2
Radiculopathy (Nervous system disorders) | 1 | 2
Seizure Disorder (Nervous system disorders) | 2 | 0
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 6 | 11
Spells (Nervous system disorders) | 1 | 1
Subarachnoid Hemorrhage (Nervous system disorders) | 0 | 2
Subdural Haemorrhage (Nervous system disorders) | 2 | 3
Transient Global Amnesia (Nervous system disorders) | 2 | 0
Transient Ischemic Attack (TIA) (Nervous system disorders) | 16 | 19
Vertigo (Nervous system disorders) | 3 | 3
Device Embolization (Product Issues) | 6 | 2
Device Malposition or Malfunction (Product Issues) | 1 | 8
Thrombus on Device (Product Issues) | 1 | 1
Suicide (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 2 | 0
Acute Renal Failure (Renal and urinary disorders) | 0 | 1
Kidney Cyst (Renal and urinary disorders) | 1 | 0
Phimosis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 3 | 3
Acute Kidney Injury (Renal and urinary disorders) | 9 | 7
Chronic Renal Failure (Renal and urinary disorders) | 3 | 3
Cystitis (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 17 | 12
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Infarct (Renal and urinary disorders) | 0 | 1
Urinary Calculi (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 2
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 15 | 28
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Residual Shunt Requiring Closure (Surgical and medical procedures) | 1 | 1
Surgical Closure of ASD (Surgical and medical procedures) | 1 | 1
Claudication (Vascular disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 1 | 0
Seroma (Vascular disorders) | 1 | 0
Vascular Ischemia (Vascular disorders) | 2 | 0
Abdominal Bleeding (Vascular disorders) | 1 | 0
Arterial Hypertension/Hypertension (Vascular disorders) | 2 | 4
Bleeding (Vascular disorders) | 10 | 15
Blood Loss (Vascular disorders) | 2 | 2
Carotid Stenosis (Vascular disorders) | 4 | 0
Deep Vein/Venous Thrombosis (Vascular disorders) | 7 | 7
Epistaxis (Vascular disorders) | 13 | 4
Hematoma (Vascular disorders) | 8 | 13
Hemoptysis (Vascular disorders) | 3 | 3
Hypotension (Vascular disorders) | 8 | 7
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusion (Vascular disorders) | 4 | 3
Peripheral Vascular Disease (Vascular disorders) | 8 | 5
Peripheral Venous Thrombus (Vascular disorders) | 1 | 1
Syncope (Vascular disorders) | 16 | 17
Systemic Embolism (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amulet (N=934) | WATCHMAN (Control) (N=944)
Abdominal Bloating (Vascular disorders) | 1 | 0
Abnormal Lab Value (Investigations) | 2 | 0
Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 3
Air Embolus (Injury, poisoning and procedural complications) | 1 | 1
Allergic Drug Reaction (General disorders) | 0 | 1
Allergic Dye Reaction (General disorders) | 1 | 0
Anemias (Blood and lymphatic system disorders) | 16 | 10
Angina Pectoris (Cardiac disorders) | 0 | 1
Aortic Valve Stenosis (Cardiac disorders) | 1 | 0
Arm Fracture (Injury, poisoning and procedural complications) | 0 | 1
Arm Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arterial Hypertension/Hypertension (Vascular disorders) | 1 | 1
Arteriovenous Malformation (Vascular disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 5
Atrial Flutter (Cardiac disorders) | 0 | 1
Bacteremia (Infections and infestations) | 2 | 0
Bleeding (Vascular disorders) | 18 | 12
Blood Loss (Vascular disorders) | 1 | 0
Blurred Vision (Nervous system disorders) | 1 | 0
Borderline Prolongation of QT Interval (Cardiac disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bruise/Purpura Simplex (Skin and subcutaneous tissue disorders) | 26 | 22
Cardiac Thrombus (Cardiac disorders) | 14 | 13
Carotid Stenosis (Vascular disorders) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 4
Chest Pain (Cardiac disorders) | 6 | 2
Cognitive Impairment (Nervous system disorders) | 1 | 0
Confusion (Nervous system disorders) | 3 | 2
Congestive Heart Failure (Cardiac disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Decreased Left Ventricular (LV) Function (Cardiac disorders) | 0 | 1
Deep Vein/Venous Thrombosis (Vascular disorders) | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Device Malposition or Malfunction (Product Issues) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Diastolic Dysfunction (Cardiac disorders) | 1 | 0
Diplopia/Double Vision (Nervous system disorders) | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Dysarthria/Slurred Speech (Nervous system disorders) | 2 | 1
Dyspnea (Cardiac disorders) | 4 | 2
Echo Finding (Investigations) | 1 | 0
Edema (Metabolism and nutrition disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 4
Epistaxis (Vascular disorders) | 37 | 33
Eye Bleed (Vascular disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 8 | 1
Fatigue/Generalized Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Fungal Infections (Infections and infestations) | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 29 | 37
Gingival Bleeding (Gastrointestinal disorders) | 2 | 1
Hemarthrosis (Vascular disorders) | 0 | 2
Hematemesis (Gastrointestinal disorders) | 0 | 1
Hematoma (Vascular disorders) | 6 | 5
Hematuria (Renal and urinary disorders) | 22 | 22
Hemoptysis (Vascular disorders) | 3 | 3
Hemorrhage (Nervous system disorders) | 0 | 1
Hemothorax (Injury, poisoning and procedural complications) | 1 | 0
Hepatic and Biliary Disorders (Hepatobiliary disorders) | 1 | 0
Hypertensive Crisis (Cardiac disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 5
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Iron-Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 1
Lacerations (Injury, poisoning and procedural complications) | 6 | 9
Lightheadedness (Vascular disorders) | 1 | 0
Loss of Speech/Stuttering (Nervous system disorders) | 0 | 1
Macular Edema (Eye disorders) | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Memory Difficulty (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 2 | 0
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 0 | 1
Mitral Valve Stenosis (Cardiac disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Neck Pain (General disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
New and Different Onset of Migraine Symptoms (Nervous system disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Numbness (Nervous system disorders) | 0 | 1
Other (General disorders) | 3 | 4
Pain (General disorders) | 0 | 1
Paresthesia/Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 0 | 2
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 0 | 1
Patent Foramen Ovale (PFO) (Cardiac disorders) | 3 | 1
Pericardial Effusion (Cardiac disorders) | 20 | 15
Pericarditis (Cardiac disorders) | 1 | 0
Peripheral Vascular Disease (Vascular disorders) | 1 | 1
Peripheral Venous Thrombus (Vascular disorders) | 3 | 1
Phlebitis (Infections and infestations) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pneumonia (Infections and infestations) | 0 | 1
Pruritis/Itching (Skin and subcutaneous tissue disorders) | 0 | 1
Residual Shunt (Surgical and medical procedures) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ST Segment Changes (Investigations) | 0 | 1
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 1 | 0
Skin Bruise (Skin and subcutaneous tissue disorders) | 3 | 4
Skin Lesions (Skin and subcutaneous tissue disorders) | 0 | 1
Sore Throat (General disorders) | 0 | 1
Spells (Nervous system disorders) | 4 | 12
Subdural Haemorrhage (Nervous system disorders) | 0 | 1
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Syncope (Vascular disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombus on Device (Product Issues) | 2 | 3
Transient Global Amnesia (Nervous system disorders) | 1 | 0
Transient Ischemic Attack (TIA) (Nervous system disorders) | 7 | 4
Trauma (Injury, poisoning and procedural complications) | 8 | 3
Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation: Tricuspid Valve (Cardiac disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 3 | 3
Urinary Tract Infections (Renal and urinary disorders) | 8 | 2
VASC AV Fistula (Cardiac disorders) | 0 | 1
VASC Bleeding (Injury, poisoning and procedural complications) | 13 | 12
VASC Bruise (Injury, poisoning and procedural complications) | 3 | 0
VASC Hematoma (Injury, poisoning and procedural complications) | 13 | 19
VASC Pain (Injury, poisoning and procedural complications) | 1 | 1
VASC Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Weakness (General disorders) | 3 | 1
Wenckebach (Mobitz I) Block (Cardiac disorders) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02879448/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02879448/SAP_001.pdf